CLINICAL TRIAL: NCT02813603
Title: Comparison of the Diagnostic Yield Between Various Endobronchial Ultrasound-guided-transbronchial Needles (EBUS-TBN) to Evaluate Suspect Mediastinal and Hilar Lymph Nodes
Brief Title: Comparison of 22-gauge and 19-gauge Aspiration Needle During EBUS-TBNA
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, Kaid Darwiche, Priv. Doz. Dr. med. Kaid Darwiche, University Hospital, Essen
Other Study IDs: EBUS19VS22
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: EBUS-TBNA; staging; lymph node metastases
MeSH Terms: conditions — Lung Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study Product (19-gauge): After randomization, the subject undergo EBUS-TBNA either with the 19-gauge needle or the 22-gauge needle
  Interventions: Procedure: EBUS
- Control Intervention (22-gauge): After randomization, the subject undergo EBUS-TBNA either with the 19-gauge needle or the 22-gauge needle
  Interventions: Procedure: EBUS

INTERVENTIONS:
Procedure: EBUS — 19G and 22G EBUS needles are compared in a randomized prospective way in lung cancer patients with enlarged mediastinal lymph nodes.

SUMMARY:
Investigators intend to compare the 19-gauge needle and the 22-gauge-needle during EBUS-TBNA concerning the diagnostic yield, the quality and quantity of each biopsy needle without raising the rate of complications.

DETAILED DESCRIPTION:
Investigators intend to compare the 19-gauge needle and the 22-gauge-needle during EBUS-TBNA performed in rigid bronchoscopy for patients with probable lung cancer diagnosis and enlarged mediastinal lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged over 18
* Patients signed written informed consent
* Mediastinal or hilar enlarged lymph nodes (>10mm) in short axis radiological or clinical findings likely for lung cancer

Exclusion Criteria:

* Severe impairment of any organs, with do not enable anaesthesia
* Quick <80%, INR >1,5, thrombocytes <50/nl or PTT>120sec
* Other clinically relevant medical or psychological diseases, which affect the patients judgement or ability to participate in this study.
* Insufficient language ability (spoken and written German)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 Patients with lung cancer and enlarged lymph nodes will be included in this study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
sample weight | February 2017

SECONDARY OUTCOMES:
The number of complications like bleeding, infections, pneumothorax and pain | February 2017

CONTACTS AND LOCATIONS:
Overall Officials: Kaid Darwiche, PD Dr. med., Study Director — supervising doctor
Locations (2):
- Ruhrlandklinik, University Hospital Essen, Essen, North Rhine-Westphalia, Germany
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolters C, Darwiche K, Franzen D, Hager T, Bode-Lesnievska B, Kneuertz PJ, He K, Koenig M, Freitag L, Wei L, Eisenmann S, Taube C, Weinreich G, Oezkan F. A Prospective, Randomized Trial for the Comparison of 19-G and 22-G Endobronchial Ultrasound-Guided Transbronchial Aspiration Needles; Introducing a Novel End Point of Sample Weight Corrected for Blood Content. Clin Lung Cancer. 2019 May;20(3):e265-e273. doi: 10.1016/j.cllc.2019.02.019. Epub 2019 Mar 4. PMID 30914312